CLINICAL TRIAL: NCT07340658
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Phase III Study to Evaluate the Efficacy and Safety of Letrozole SIE Compared to Femara® (Both in Combination With the CDK4/6 Inhibitor Palbociclib) in Postmenopausal Women With HR-Positive, HER2-Negative, Inoperable Locally Advanced or Metastatic Breast Cancer (SIE-3)
Brief Title: A Study to Investigate the Efficacy and Safety of Letrozole SIE Compared With Femara® (Both Combined With the CDK4/6 Inhibitor Palbociclib) in Postmenopausal Women With HR-Positive, HER2-Negative, Advanced Breast Cancer
Acronym: SIE-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROV-SIE-2025-02; 2025-524846-85-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced, Metastatic Breast Cancer
Keywords: Letrozole SIE; Advanced breast cancer; Metastatic breast cancer; Endocrine therapy; Efficacy; Safety; Palbociclib; Injectable
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole SIE (Experimental)
  Interventions: Drug: Letrozole SIE + Palbociclib + Oral placebo
- Femara® 2.5 mg (Active Comparator)
  Interventions: Drug: Oral Femara® + Palbociclib + Injectable placebo

INTERVENTIONS:
Drug: Letrozole SIE + Palbociclib + Oral placebo — Letrozole SIE quarterly (injectable) + Palbociclib once daily (oral) + placebo once daily (oral)
  Arms: Letrozole SIE
Drug: Oral Femara® + Palbociclib + Injectable placebo — Femara® 2.5 mg/day (oral) + Palbociclib once daily (oral) + placebo quarterly (injectable)
  Arms: Femara® 2.5 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Letrozole SIE (injectable) compared to Femara® (oral tablet), both given together with palbociclib, for the first-line treatment of postmenopausal women with HR-positive, HER2-negative, inoperable locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, active-controlled Phase III study comparing Letrozole SIE with Femara® (both in combination with the CDK4/6 inhibitor palbociclib) in postmenopausal women with HR-positive, HER2-negative, inoperable locally advanced or metastatic breast cancer. The study employs double-blinding with matching placebos (double-dummy technique) to minimize bias on the part of participants, investigators, and analysts. Participants will be randomized in a 1:1 ratio to receive either Letrozole SIE (experimental use) or Femara® (active comparator), both in combination with the CDK4/6 inhibitor palbociclib. Randomization occurs after Screening and confirmation of eligibility and will be stratified by visceral metastasis (Yes/No) and prior adjuvant endocrine therapy (Yes/No).

The Treatment Period will last from Cycle 1 Day 1 (C1D1) until study intervention discontinuation due to disease progression, symptomatic deterioration, unacceptable toxicity, withdrawal of consent, loss to follow-up, participant's death, or end of study, whichever occurs first. After study intervention discontinuation, a post-discontinuation visit will be performed. Then, participants will be followed until withdrawal of consent, loss to follow-up, the participant's death, or end of study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with inoperable locally advanced or metastatic breast cancer.
* Confirmed diagnosis of HR-positive/HER2-negative breast cancer.
* Postmenopausal woman.
* Previously untreated with any systemic anticancer therapy for their locoregionally recurrent or metastatic HR-positive disease. Participants may have received cytotoxic chemotherapy within (neo) adjuvant previous treatment of breast cancer but must show progressive disease prior to enrolment.
* Have either measurable disease or non-measurable bone-only disease.
* ECOG performance status 0-2.
* Adequate organ and marrow function.
* Resolution of all acute toxic effects of prior anticancer therapy or surgical procedures to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the participant at the investigator's discretion).
* BMI ≥ 19 and ≤ 39 kg/m2.

Exclusion Criteria:

* Participants with advanced, symptomatic, visceral spread who are at risk of life-threatening complications in the short term.
* Known uncontrolled or symptomatic central nervous system (CNS) metastases.
* Concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer.
* Active cardiac disease or a history of cardiac dysfunction.
* Uncontrolled hypertension.
* History of symptomatic vertebral fragility fracture or any fragility fracture of the hip, pelvis, wrist, or other location (defined as any fracture without a history of trauma or because of a fall from standing height or less, excluding fingers, toes, face and skull).
* Presence of medical conditions associated with low bone mass.
* Presence of detectable viral infection, including HBV, HCV, and HIV. Screening is not required for enrollment. Note: Participants who have been effectively treated and have a sustained virologic response are eligible for enrollment.
* Major surgery, chemotherapy, radiotherapy, any investigational agents, or other anticancer therapy within 14 days (2 weeks) before randomization. Participants who received prior radiotherapy to > 25% of bone marrow are not eligible independent of when it was received.
* Bisphosphonates or receptor activator of nuclear factor kappa-β ligand (RANKL) inhibitors initiated or have their dose changed within 14 days prior to randomization, i.e., participants should be on stable dose treatment for at least 14 days prior to randomization.
* Use of estrogen or progesterone hormone replacement therapy, oral contraceptives, androgens, LHRH analogs, prolactin inhibitors, or antiandrogens within 3 months prior to randomization.
* Use of the following medications within the three previous days or a period of 5 half-lives, whichever is longer prior to randomization:

  1. Any medications including St. John's wort, known to be potent or moderate inducers of Cytochrome P450 (CYP) 3A.
  2. Any medications or products known to be potent or moderate inhibitors of CYP3A (e.g., grapefruit juice).
  3. Any medications known to be inducers of CYP2A6.
  4. Any medications known to be inhibitors of CYP2A6.
* Concurrently use of other anticancer therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From the date of randomization to the date of the first documented progression or death due to any cause, assessed according to RECIST version 1.1 (up to approximately 32 months).
  PFS per Investigator assessment, defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS will be assessed via a local radiology assessment according to RECIST v1.1. PFS as assessed through a blinded independent central review will be used for supportive evidence of the primary efficacy endpoint.

SECONDARY OUTCOMES:
Overall Survival (OS): Primary analysis | From the date of randomization to date of death from any cause (up to approximately 32 months).
  OS, defined as the time from the date of randomization to date of death from any cause.
Overall Survival (OS): Final analysis | From the date of randomization to date of death from any cause (up to approximately 60 months).
  OS, defined as the time from the date of randomization to date of death from any cause.
Objective Response Rate (ORR): Primary analysis | From the date of randomization to the date of the first documented progression or death due to any cause, assessed according to RECIST version 1.1 (up to approximately 32 months).
  ORR, defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) by Investigator assessment per RECIST v1.1 criteria.
Objective Response Rate (ORR): Final analysis | From the date of randomization to the date of the first documented progression or death due to any cause, assessed according to RECIST version 1.1 (up to approximately 60 months).
  ORR, defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) by Investigator assessment per RECIST v1.1 criteria.
Incidence of arthralgias/arthritis and/or myalgias | From the date of the first dose of study intervention to the post-discontinuation visit (up to approximately 32 months).
  To compare the incidence rate of a combined event of arthralgias/arthritis and/or myalgias between Letrozole SIE and Femara®
Time to Response (TTR) | From the date of randomization to the date of the first documented evidence of complete response or partial response (up to approximately 32 months).
  TTR, defined for participants with complete response or partial response defined by Investigator assessment per RECIST v1.1 criteria as the interval between randomization and the earliest documentation of response.
Duration of response (DOR) | From first documented evidence of complete response (CR) or partial response (PR) until disease progression or death from any cause, whichever occurs first (up to approximately 32 months).
  DOR, defined for those participants with complete response (CR) or partial response (PR) as the time from first documented evidence of CR or PR until disease progression by Investigator assessment per RECIST v1.1 criteria, or death from any cause, whichever occurs first.
Clinical benefit rate (CBR) | From the date of randomization to the date of the first documented progression or death due to any cause, assessed according to RECIST version 1.1 (up to approximately 32 months).
  CBR, defined as the proportion of participants with complete response (CR), partial response (PR), or stable disease (SD) ≥ 6 months according to Investigator assessment per RECIST v1.1 criteria
Time to treatment failure (TTF) | From date of randomization to study intervention discontinuation for any reason (up to approximately 32 months).
  TTF, defined as the time from randomization to study intervention discontinuation for any reason.
Change from baseline in the FACT-G total score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-G questionnaire. FACT is a modular approach to assess participant health-related quality of life using a 'core' set of questions (FACT-G) as well as a cancer site-specific module. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. For all questions, participants are asked to respond to a five-level scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
Change from baseline in the FACT-G Physical well-being subscale score | From the date of randomization to the time of disease progression (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-G subscales.
Change from baseline in the FACT-G Social/Familiy well-being subscale score | From the date of randomization to the time of disease progression (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-G subscales.
Change from baseline in the FACT-G Emotional well-being subscale score | From the date of randomization to the time of disease progression (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-G subscales.
Change from baseline in the FACT-G Functional well-being subscale score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-G subscales.
Change from baseline in the FACT-B total score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using FACT-B questionnaire. FACT is a modular approach to assess participant health-related quality of life using a 'core' set of questions (FACT-G) as well as a cancer site-specific module. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The FACT-B consists of the FACT-G and a breast-specific module: a 10-item instrument designed to assess participant concerns relating to breast cancer. For all questions, participants were asked to respond to a five-level scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
Change from baseline in the FACT-B Breast Cancer subscale score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using the FACT-B questionnaire.
Change from baseline in the FACT-ES total score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using the FACT-ES questionnaire. FACT is a modular approach to assess participant health-related quality of life using a 'core' set of questions (FACT-G) as well as a cancer site-specific module. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. FACT-ES incorporates 19 additional items that assess endocrine related symptoms in addition to the FACT-G core items. For all questions, participants were asked to respond to a five-level scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
Change from baseline in the FACT-ES Endocrine Symptoms subscale score | From the date of randomization to the post-discontinuation visit (up to approximately 32 months).
  To compare the health-related quality of life between Letrozole SIE and Femara® (both in combination with the CDK4/6 inhibitor palbociclib) using the FACT-ES questionnaire.
Time to deterioration in the FACT-G total score | From the date of randomization to to the first occurrence of a decrease from baseline of at least 5 points for FACT-G (up to approximately 32 months).
  Deterioration will be defined as the time from the date of randomization to the first occurrence of a decrease from baseline of at least 5 points for FACT-G total score.
Time to deterioration in the FACT-B total score | From the date of randomization to to the first occurrence of a decrease from baseline of at least 7 points for FACT-B (up to approximately 32 months).
  Deterioration will be defined as the time from the date of randomization to the first occurrence of a decrease from baseline of at least 7 points for FACT-B total score.
Time to deterioration in the FACT-ES total score | From the date of randomization to to the first occurrence of a decrease from baseline of at least 7 points for FACT-ES (up to approximately 32 months).
  Deterioration will be defined as the time from the date of randomization to the first occurrence of a decrease from baseline of at least 7 points for FACT-ES total score.
ESR1 mutation status | From the date of randomization to the time of disease progression (up to approximately 32 months).
  Percentage of participants with ESR1 mutations at the time of disease progression among those without ESR1 mutations at baseline.
ESR1 mutant allele frequency | At the time of disease progression (up to approximately 32 months).
  ESR1 mutant allele frequency at the time of disease progression.
Incidence of Adverse Events (AEs) | From the Informed Consent Form signature to the post-discontinuation visit (approximately up to 60 months).
  AEs type, severity, seriousness, and relationship to study intervention, including the incidence of TEAEs, the incidence of serious TEAEs, and the incidence of TEAEs leading to study intervention discontinuation.
Incidence of injection site reactions | From the date of the first dose of study intervention to the post-discontinuation visit (approximately up to 60 months).
  Injection site redness, swelling, and induration will be evaluated before and after Letrozole SIE or injectable placebo administration.
Changes in injection-related pain score | From the date of the first dose of study intervention to the post-discontinuation visit (approximately up to 60 months).
  Injection site pain, self-assessed by participants using an numeric rating scale (NRS) at the time of Letrozole SIE or injectable placebo administration and for a longer period of time if necessary. The numeric rating scale (NRS) evaluates the intensity of injection-related pain experienced at the time of Letrozole SIE/injectable placebo administration. It is scored from 0 to 10 (0 meaning no pain and 10 meaning the worst possible pain).
Change from baseline in Bone mineral density (BMD) | From the Informed Consent Form signature to the post-discontinuation visit (approximately up to 32 months).
  Change from baseline in BMD assessed by DXA